CLINICAL TRIAL: NCT00682903
Title: Use of a Bearable Continuous Interstitial Glucose Monitoring Device (GuardianR) During Teaching Sessions to Functional Insulin Therapy Concept in Patients Suffering From Type 1 Diabetes: Evaluation at 6 and 12 Months
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/24
Record Dates: First submitted 2008-03-05; First posted 2008-05-23 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Complications
Keywords: glucose; diabetes; glycemia
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): This arm will benefit from the nonstop measure of the subcutaneous glucose during the hospitalization and the week on returning to the place of residence,
  Interventions: Device: GuardianR

INTERVENTIONS:
Device: GuardianR — As self monitoring of capillary glucose level is needed to validate those algorithms, we postulate that using a device able to permanently control interstitial glucose readable by both medical team and patient himself (during the session and the 5 following days after discharge) could significantly improve safety and efficiency of such educative session.

SUMMARY:
The objective of the project is to evaluate advantages from the use of a bearable continuous interstitial glucose monitoring device (GuardianR) during educative sessions of diabetic patients dedicated to functional insulin therapy teaching. This concept of intensified treatment is based on testing and explanation of simplified decision making algorithms to adapt insulin dose to every true life conditions. As self monitoring of capillary glucose level is needed to validate those algorithms, we postulate that using a device able to permanently control interstitial glucose readable by both medical team and patient himself (during the session and the 5 following days after discharge) could significantly improve safety and efficiency of such educative session.

DETAILED DESCRIPTION:
Two groups of 60 patients (experimental and control groups) will be followed and evaluated at 6 and 12 months. We do think that this new tool would facilitate education of patients and lead further to a better glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Subject major, from 18 to 70 years old
* Diabetes of type 1 defined according to the criteria of American Diabetes Association
* Insulinic treatment for at least 12 months
* Understood HbA1C enters 6,5 and 9,5 %

Exclusion Criteria:

* Minor subjects or under guardianship
* Unbalance kétosis current or recent
* Pregnancy
* Incapacitated to participate weekly complete educational in the functional insulin-therapy,
* Evolutionary severe general disease
* Psychiatric confusions
* Unbalance chronic (HbA1c > 9,5 %) connected to an absence of adapted coverage or to abnormal behaviors
* Pathology making not interpretable the rate of HbA1c (hemoglobinopathy, anemia)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The HbA1c, the witness of the quality of the metabolic balance, in 6 and 12 months. We shall compare the deltae of HbA1c between the period of inclusion and 6 and 12 months following the training course in the "fonctional" insulin therapy | glycemia

CONTACTS AND LOCATIONS:
Locations (1):
- CHU timone, Marseille, Bouches du Rhone, France